CLINICAL TRIAL: NCT05512299
Title: Investigating Cerebellar Inhibition and Its Clinical Significance in Parkinsonian Tremor and Intention Tremor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: CMUH111-REC3-014
Record Dates: First submitted 2022-08-19; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Tremor
Keywords: cerebellar inhibition; pallidothalamic tractotomy; thalamotomy; Parkinson's disease; MR-guided focused ultrasound
MeSH Terms: conditions — Tremor; Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PD with resting tremor: Parkinson's disease patient with pure resting tremor.
  Interventions: Diagnostic Test: Transcranial Magnetic Stimulation
- PD with postural tremor: Parkinson's disease patient with postural tremor.
  Interventions: Diagnostic Test: Transcranial Magnetic Stimulation
- Cerebellar degeneration with intention tremor: Cerebellar degeneration patient with intention tremor.
  Interventions: Diagnostic Test: Transcranial Magnetic Stimulation

INTERVENTIONS:
Diagnostic Test: Transcranial Magnetic Stimulation — The CBI is recorded with two different TMS coils. The figure-of-eight coil (2X90 mm) is used for the motor cortex stimulation and the double cone coil (2X126 mm) is used for the cerebellar stimulation. The target recording muscle is first dorsal interosseous (FDI). The TMS intensity used to induce an average MEP amplitude of 0.5 mV is also determined. CBI is measured by a paired TMS with an inter-stimulus interval of 6 ms. That is, the test TMS at M1 is delivered 6 ms following the conditional TMS at contralateral cerebellum.

SUMMARY:
Cerebellocerebral connection plays an important function in motor control. Nowadays it can be investigated with neuroimaging and physiological methods in humans. Cerebellar inhibition (CBI) is a phenomenon showing a physiological suppression of the motor evoked potential (MEP) evoked from the motor cortex (M1) by delivering a preceding transcranial magnetic stimulation (TMS) on the contralateral cerebellum. Despite the mediated pathway is supposed to be the cerebello-dentato-thalamo-cortical (CDTC) circuit, there is no conclusive evidence. In addition, the clinical significant of CBI remains unclear. Based on our previous studies, we found that the patients with advanced tremor show an impaired Bereitschaftspotential. The findings support a notion that the patients with tremor bear dysfunction of the CDTC circuit. Intriguingly, the pathogenesis of the parkinsonian tremor is highly associated with the CDTC circuit. The "dimmer-switch" model suggests that the basal ganglia-thalamo-cortical circuit dysfunction may initiate the resting tremor, and the following CDTC circuit dysfunction will lead to the large-amplitude resting and postural tremor in Parkinson's disease (PD). The intention tremor is usually found in the patients with cerebellar degeneration, which is also relevant to the CDTC circuit dysfunction. We expect that the clinical significance of CBI and the mediated pathway of CBI will be clarified by this study.

DETAILED DESCRIPTION:
The patients with hereditary cerebellar degeneration usually present intention tremor. Whether the intention tremor and the other cerebellar signs are correlated with their CBI finding remains unclear. By measuring the excitability curve (or input-output curve) of the CBI, we will be able to clarify this issue.

We will first examine the relationship between CBI and clinical manifestations, particularly the different tremor types. Any CBI change following the PTT intervention in the PD patients will provide an excellent opportunity to investigate the relevance of the basal ganglia-thalamo-cortical circuit with CBI. The DTI findings will provide additional support to our hypothesis.

In the first part of the study, we will recruit twenty age-matched patients into the three groups: PD with pure resting tremor, PD with postural tremor and cerebellar degeneration with intention tremor. They will receive clinical assessments, deep phenotyping with eye tracking, tremor recording and gait analysis. Diffusion tensor imaging focusing on pallidothalamic and dentatothalamic tractography will be done. The excitability curve of CBI will be examined with five TMS intensity steps. We suppose that there will be a gradient correlation of the CBI with the three tremor groups and the two diffusion tensor imaging tracts. In the second part of the study, we will follow up the PD patients who receive the pallidothalamic tractotomy via magnetic resonance imaging-guided focus ultrasound (MRg-FUS). Twelve PD patients with pure resting tremor and twelve PD patients with postural tremor will be monitored for one year. The pallidothalamic tractotomy provides an excellent opportunity to verify our findings in the first part. We suppose that the CBI change will occur in the patients with postural tremor instead of those with pure resting tremor. In summary, we expect that the clinical significance of CBI and the mediated pathway of CBI will be clarified by this study.

ELIGIBILITY:
Inclusion Criteria:

Patients meet the diagnosis of PD with resting/postural or cerebellar degeneration with intention tremor based on the established consensus criteria.

Exclusion Criteria:

1. Patients with contraindication to TMS or MRI examination.
2. Impairment of cognition that leads unable to fully cooperate with the oral commands during examinations.
3. Functional III or above congestive heart failure, or cancer with distant metastasis.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult PD patients with pure resting tremor or mixed resting and postural tremor will be studied. Some of them are the patients receiving MR-guided focus ultrasound (MRgFUS). In addition, patients with cerebellar degeneration with intention tremor will be also recruited. Those patients with contraindication to TMS or MRI examination will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline cerebellar inhibition (CBI) input output curve | baseline (before the MRgFUS), 1-day, 24-weeks and 48-weeks after the MRgFUS
  The CBI is recorded with two different TMS coils. The figure-of-eight coil (2X90 mm) is used for the motor cortex stimulation and the double cone coil (2X126 mm) is used for the cerebellar stimulation. The target recording muscle is first dorsal interosseous (FDI). The TMS intensity used to induce an average MEP amplitude of 0.5 mV is also determined. CBI is measured by a paired TMS with an inter-stimulus interval of 6 ms. That is, the test TMS at M1 is delivered 6 ms following the conditional TMS at contralateral cerebellum.
  There are five TMS intensities used for the conditional cerebellar stimulation: 80%, 90%, 100%, 110% and 120% inion active motor threshold. Ten trials are recorded for each TMS intensity with a pseudorandomized order. The interval between two cerebellum-M1 TMS pairs is 8-seconds with 25% variability (i.e. 6-10 s) to reduce the prediction bias.
Change from baseline functional magnetic resonance imaging | baseline (before the MRgFUS), 48-weeks after the MRgFUS
  In this study we mainly adopt diffusion tensor imaging (DTI) to quantify two interested projections: the pallidothalamic pathway and the dentatothalamic pathway.
  Diffusion tensor imaging of fifty gradient directions is acquired with five non-gradient (B0) images. The B-value is 1500 s/mm2, FOV = 240mm x 240mm, image matrix = 96 x 96, slice thickness = 2.5mm with zero gap. The voxel size is 2.5 x 2.5 x 2.5 mm3 isotopically. The TR was approximately 10000ms which is adjusted to match the slice number of requirements. Image acquired with axial direction, 56 slices to cover the whole brain.

SECONDARY OUTCOMES:
Change from baseline clinical evaluations | baseline (before the MRgFUS), 1-day, 24-weeks and 48-weeks after the MRgFUS
  In addition to a detailed history and neurological examinations, the clinical assessment also includes International Parkinson and Movement Disorder Society-sponsored UPDRS (MDS-UPDRS) and clinical rating scale for tremor (CRST)for the PD patients. The Scale for the Assessment and Rating of Ataxia (SARA) and CRST are adopted for the patients with cerebellar degeneration.
Change from baseline gait analysis | baseline (before the MRgFUS), 1-day, 24-weeks and 48-weeks after the MRgFUS
  The gait analysis system (Zeno Walkway System with PKMAS) provides detailed gait parameters including velocity, cadence, pressure and cyclogram.
  Variables in gait analysis: 1.Gait initiation, 2.Level walking, 3.Gait termination.
Change from baseline surface electromyography and eye-tracking pattern | baseline (before the MRgFUS), 1-day, 24-weeks and 48-weeks after the MRgFUS
  The pattern of eye-tracking and surface electromyography (SEMG) with accelerometer will be recorded to monitor the therapy outcome. The eye-tracking system (EyeLink 1000 Plus) will track eye movements regarding the target fixation, saccade, smooth pursuit and image stimuli. The multiple SEMG recording (CED Power1401) will focus on the arm and hand muscles relevant to the tremor (e.g. first dorsal interosseous, abductor pollicis brevis, extensor carpi radialis and flexor carpi radialis). The accelerometer can also reveal the mechanical information of the tremor oscillation.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Kuei Lu, MD, PhD, Principal Investigator — Department of Neurology, China Medical University Hospital
Locations (1):
- Department of Neurology, China Medical University Hospital, Taichung, Taiwan